CLINICAL TRIAL: NCT02458053
Title: Testing the Efficacy of a Spousal Support Enhanced Weight Loss Program on Weight Loss Among African American Men
Acronym: TEAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-3193
Record Dates: First submitted 2015-05-27; First posted 2015-05-29 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Overweight; Weight Loss; Obese
Keywords: African American; male; couples; randomized control trial
MeSH Terms: conditions — Overweight; Weight Loss; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TEAM Enhanced (Experimental): The enhanced intervention will include group sessions where the participant attends with partner ( including a couples skill training session), weekly tailored feedback, and weekly lessons.
  Interventions: Behavioral: Attends with partner; Behavioral: Couples Skill Training; Behavioral: Face to face group sessions; Behavioral: Self Monitor; Other: Notebook; Behavioral: Feedback
- TEAM Traditional (Active Comparator): The intervention will include group sessions where the male attends alone, weekly tailored feedback, and weekly lessons.
  Interventions: Behavioral: Face to face group sessions; Behavioral: Self Monitor; Other: Notebook; Behavioral: Feedback

INTERVENTIONS:
Behavioral: Attends with partner — The index partner will participate in intervention as a couple with their female counterpart.
  Arms: TEAM Enhanced
Behavioral: Couples Skill Training — Participants and their partners will attend a pre session covering topics to assist them in working together to facilitate lifestyle changes.
  Arms: TEAM Enhanced
Behavioral: Face to face group sessions — Group sessions will consists of components in traditional weight management programs.
Behavioral: Self Monitor — Participants will be instructed to monitor their eating and physical activity behaviors online/mobile application.
Other: Notebook — The notebook will consist of behavioral lessons, diet and physical activity plans, and additional resources to assist participants in achieving their behavioral goals.
Behavioral: Feedback — Each participant will receive a tailored email providing feedback on their weekly progress.

SUMMARY:
The purpose of this study is to determine the effect of a spousal support enhanced weight loss program on weight loss among African American men.

DETAILED DESCRIPTION:
In 2012, African Americans (AA) were 1.4 times more likely to be overweight and obese than non-Hispanic Whites. The Office of Minority Health reports the prevalence of overweight and obesity (BMI>25) among AA men age 20 and older is 70%. AA men suffer disproportionately from obesity-related consequences. Modest weight loss (WL) of 10% or less improves cardiovascular disease risk factors and reduces the risk of type 2 diabetes. However, the majority of participants in lifestyle weight loss (LWL) interventions are most commonly Caucasian women. While men are unrepresented in weight loss programs; even fewer studies examine WL in AA men. Only 4.5% of AA men participate in research studies, according to the National Institute of Health (NIH). When AA men have participated in LWL interventions, they have loss less weight compared to Caucasian men. Consequently, the evidence on the appropriateness of the current WL strategies and recommendations for AA men is limited.

There is limited literature on the appropriate strategies for WL in AA men because of their lack of participation. Social support is a predictor of weight loss and support from family is important in AA culture. Spousal support results, defined as spouse or significant other, are inconsistent and are largely conducted in Caucasian populations. The use of individual based theoretical frameworks may explain these inconsistencies. Using a dyad based framework like the Interdependence Theory may produce different results. The use of a dyad based theoretical framework and testing the effects of spousal support adds to the literature of WL among AA men.

This study seeks to determine the best strategies to attract overweight and obese AA men to participate and examine the efficacy of a 3 month spousal support enhanced behavioral weight loss intervention focused on behavior modification, nutrition and physical activity compared to a traditional intervention in achieving clinical significant weight loss in AA men. Using 2 arms randomized controlled trial (RCT) 26 AA men and their partners will be recruited to participate in each arm in Orange, Durham and Wake County, North Carolina. The investigator hypothesizes the proposed TEAM (Together Eating & Activity Matters) program, a spousal support enhanced WL intervention, will result in clinical weight loss among AA men.

ELIGIBILITY:
Inclusion Criteria:

* The participant self-identifies as African American male.
* The participant is between the ages of 18 and 65.
* The participant has a BMI between 25 and 45 kg/m2.
* The participant enrolls with an African American overweight female spouse or cohabiting intimate partner
* The participant has weekly access to the internet and/or a mobile phone with internet capabilities.

Exclusion Criteria:

* Both the participant and the partner are not willing and interested in losing weight.
* The participant is taking any medications that affect weight.
* The participant is participating in any other weight loss program.
* The participant has recently lost 10 lbs or more.
* The participant is expecting to relocate within the next 6 months.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2016-02; Primary Completion 2016-12 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Weight | Baseline, 6 weeks, 12 weeks
  Body weight(kg) expressed as a continuous variable will be collected on a digital scale.

SECONDARY OUTCOMES:
Waist Circumference | Baseline,12 weeks
BMI | Baseline,12 weeks
Blood pressure | Baseline, 12 weeks
  Blood pressure will be assessed using DINAMAP monitor.
Behavior | Baseline, 12 weeks
  Changes in behavior will be assessed (e.g. diet (caloric Intake), and physical activity).
Psychosocial variables | Baseline, 12 weeks
  Changes in psychosocial variables will be assessed (Self-regulation of eating behaviors, self-efficacy of eating behaviors and physical activity).
Social Support | Baseline, 6 weeks, 12 weeks
  Social support of eating behaviors and physical activity will be assessed.
Couple/Family Variables | Baseline, 12 weeks
  Couple/ Family Variables will be assessed (e.g. marital satisfaction, transformation of motivation/communal coping, and family communication).

CONTACTS AND LOCATIONS:
Overall Officials: Deborah F Tate, PhD, Study Chair — University of North Carolina, Chapel Hill; Candice Alick, MS, Principal Investigator — University of NC-Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Alick CL, Samuel-Hodge C, Ward D, Ammerman A, Rini C, Tate DF. Together Eating & Activity Matters (TEAM): results of a pilot randomized-clinical trial of a spousal support weight loss intervention for Black men. Obes Sci Pract. 2018 Jan 17;4(1):62-75. doi: 10.1002/osp4.142. eCollection 2018 Feb. PMID 29479466